CLINICAL TRIAL: NCT03359876
Title: Evaluation of Clinical Outcomes Among Non-valvular Atrial Fibrillation Patients With Renal Dysfunction Treated With Warfarin or Reduced Dose Rivaroxaban
Brief Title: Clinical Outcomes Among Non-valvular Atrial Fibrillation Patients With Renal Dysfunction
Acronym: CALLIPER
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19721
Record Dates: First submitted 2017-11-28; First posted 2017-12-02 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: Real-world study; Atrial fibrillation; Renal dysfunction; Rivaroxaban; Warfarin
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rivaroxaban: NVAF patients with renal dysfunction newly initiated on rivaroxaban 15 mg for stroke prevention
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Warfarin: NVAF patients with renal dysfunction newly initiated on vitamin K antagonist (warfarin) for stroke prevention
  Interventions: Drug: Warfarin sodium

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 15 mg, once daily
  Groups: Rivaroxaban
Drug: Warfarin sodium — Individually adjusted dose
  Groups: Warfarin

SUMMARY:
The objective of the study is to evaluate the effectiveness and safety of the reduced dose rivaroxaban (15 mg once daily) as compared to warfarin in non-valvular atrial fibrillation (NVAF) patients with renal dysfunction in routine clinical practice. The study has a retrospective design, and will be conducted in the US Truven Health MarketScan Commercial Claims and Medicare Supplemental Databases

ELIGIBILITY:
Inclusion Criteria:

* have to be adults (≥18 years of age)
* newly-initiated on warfarin or rivaroxaban 15 mg (index event, index drug)
* have at least 365 days of continuous medical and prescription benefits prior to the index event (baseline period)
* have at least two diagnosis codes for NVAF (on outpatient or inpatient claims, at two different days) and
* have at least one diagnosis code (inpatient or outpatient) indicating renal dysfunction in the baseline period

Exclusion Criteria:

* valvular AF (at least one inpatient diagnosis in the baseline period)
* pregnancy (inpatient or outpatient diagnosis in the baseline period)
* transient cause of AF (inpatient or outpatient diagnosis in the baseline period)
* venous thromboembolism (pulmonary embolism or deep vein thrombosis) (one inpatient or outpatient diagnosis 60 days prior to or on the index date) or
* overcame a hip or knee replacement (one inpatient diagnosis or procedure code 60 days prior to or on the index date)
* have a pharmacy claim for an oral anticoagulation (OAC) dispensation (warfarin, apixaban, dabigatran, edoxaban or rivaroxaban) in the baseline period
* receive both warfarin and rivaroxaban 15 mg on the index date
* have an end-stage kidney disease or be on dialysis (one inpatient or outpatient diagnosis or procedure code in the baseline period).

For the main analysis, patients having malignant cancers (inpatient or outpatient diagnosis in the baseline period) will be excluded. A sensitivity analysis, omitting this exclusion criterion, will be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population of this study is all the insured individuals included in the US Truven Health MarketScan Commercial Claims and Medicare Supplemental Databases.To be included in the present study, adult patients have to be diagnosed with NVAF, have renal dysfunction and be newly-initiated on warfarin or rivaroxaban 15 mg for stroke prevention.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke | Retrospective analysis from August 2011 to September 2017
  The study outcomes will be defined based on the International Classification of Diseases, 9th- and 10th-revision, Clinical Modification (ICD-9/10-CM) diagnosis codes, Current Procedural Technology, 4th-revision (CPT-4) and Healthcare Common Procedure Coding System (HCPCS) procedure codes
Intracranial hemorrhage | Retrospective analysis from August 2011 to September 2017
  The study outcomes will be defined based on ICD-9/10-CM diagnosis codes, CPT-4 and HCPCS procedure codes
Bleeding-related hospitalization | Retrospective analysis from August 2011 to September 2017
  The study outcomes will be defined based on ICD-9/10-CM diagnosis codes, CPT-4 and HCPCS procedure codes, Cunningham algorithm

SECONDARY OUTCOMES:
Composite endpoint, which is defined as the occurrence of ischemic stroke or intracranial hemorrhage | Retrospective analysis from August 2011 to September 2017
  The study outcomes will be defined based on ICD-9/10-CM diagnosis codes, CPT-4 and HCPCS procedure codes
Progression to stage 5 chronic kidney disease (CKD), kidney failure or need for dialysis | Retrospecitive analysis from August 2011 to September 2017
  The study outcomes will be defined based on ICD-9/10-CM diagnosis codes, CPT-4 and HCPCS procedure codes

CONTACTS AND LOCATIONS:
Locations (1):
- US Truven MarketScan, Whippany, New Jersey, United States

REFERENCES:
- [Derived] Vaitsiakhovich T, Coleman CI, Kleinjung F, Vardar B, Schaefer B. Worsening of kidney function in patients with atrial fibrillation and chronic kidney disease: evidence from the real-world CALLIPER study. Curr Med Res Opin. 2022 Jun;38(6):937-945. doi: 10.1080/03007995.2022.2061705. Epub 2022 Apr 22. PMID 35392744